CLINICAL TRIAL: NCT06347705
Title: Phase II Study Evaluating the Effects of Single Site Intratumoral Injections of Anti-CD40 Agonist Antibody (2141-V11) Given as Monotherapy Prior to Radical Prostatectomy to Men With Intermediate Risk Disease and in Combination With Androgen Deprivation Therapy for Those With High Risk Localized and Low Volume Metastatic Disease
Brief Title: A Study of 2141-V11 in Combination With Standard Treatments in People With Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-252
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; 2141-V11; Memorial Sloan Kettering Cancer Center; 23-352
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A (Experimental): Men presenting with clinically localized intermediate-risk disease for whom surgery can be safely delayed for neoadjuvant treatment.
  Interventions: Biological: 2141-V11 Antibody
- Cohort B (Experimental): Men presenting with clinically localized or locoregional high-risk disease.
  Interventions: Biological: 2141-V11 Antibody
- Cohort C (Experimental): Men presenting with low-volume metastatic disease for whom a multimodality therapeutic approach including removal of the primary has the potential to eliminate all disease.
  Interventions: Biological: 2141-V11 Antibody

INTERVENTIONS:
Biological: 2141-V11 Antibody — 2141-V11 Antibody: Intratumor injection

SUMMARY:
The purpose of this study is to see whether combining 2141-V11 with various standard treatments is an effective treatment approach for prostate cancer. 2141-V11 works by activating the immune system to find and kill cancer cells. Researchers will look at whether this treatment approach is able to completely get rid of cancer in participants, and they will check for the presence of minimal residual disease (MRD) in participants. MRD is a small number of cancer cells that can be detected in the body after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent and Authorization for Use and Release of Health and Research Study Information (HIPAA authorization) NOTE: HIPAA authorization may be either included in the informed consent or obtained separately
* Male aged 18 years and above
* Serum testosterone of ≥150 ng/dL (Cohorts B and C) except for patients currently on ADT.
* Adequate bone marrow, hepatic, and renal function, as evidenced within 28 days prior to treatment start by:

ANC ≥1500/µl (≥1000/µl if benign ethnic neutropenia) Hemoglobin ≥9 g/dL Platelet count ≥100,000/µl Creatinine Clearance Measure by Cockcroft-Gault Formula >45 mL/min Total Bilirubin ≤ 1.8 mg/dl (Note: In participants with Gilbert's syndrome, if total bilirubin is 1.8 mg/dL, measure direct and indirect bilirubin and if direct bilirubin is ≤1.5 × ULN, participant may be eligible) SGOT (AST) ≤ 92.5 U/L SGPT (ALT) ≤ 137 U/L

* Participants must have a clinical T stage documented by the treating urologist/medical oncologist within 90 days prior to treatment start using the 8th edition American Joint Committee on Cancer (AJCC) staging system, recorded as the urologist's/medical oncologist's best clinical assessment of extent of local disease by digital rectal examination and/or available imaging studies such as transrectal ultrasound, CT scan, and/or MRI. (Applicable to Cohorts A, B and C).
* Candidate for RP with lymph node dissection as per the investigator
* Agrees to use a condom (even men with vasectomies) and another effective method of birth control if he is having sex with a woman of childbearing potential or agrees to use a condom if he is having sex with a woman who is pregnant while on study drug and for 3 months following the last dose of study drug. Must also agree not to donate sperm during the study and for 3 months after receiving the last dose of study drug.
* Evidence of a prostate lesion on prostate magnetic resonance imaging scan

Exclusion Criteria:

Participants that meet any of the criteria listed below will not be eligible for study entry:

* Prior prostate surgery, pelvic lymph node dissection, radiation therapy, or focal therapy as a treatment for prostate cancer or benign prostatic disease.
* Current ADT with GnRH antagonist/agonist and/or ARSI initiated >12 weeks enrollment.
* Prior cytotoxic chemotherapy for prostate cancer
* Prior experimental therapy for prostate cancer within 30 days of planned Cycle 1 of 2141-V11.
* Known brain, liver, lung or other visceral metastasis (with the exception of retroperitoneal and / or pelvic nodal metastases as per inclusion criteria)
* Prior prostate cancer metastasis-directed therapies other than described above.
* Currently active second malignancy or past medical history of malignancies diagnosed within the last 5 years that require active therapy and/or in remission with life expectancy of < 5 years, with the exception of resected non-melanoma skin cancers, non-muscle invasive bladder cancer, stage I head and neck cancer, or stage I colorectal cancer.
* Significant medical condition other than cancer, that would prevent consistent and compliant participation in the study that would, in the opinion of the investigator, make this protocol unreasonably hazardous including but not limited to:

  * Any medical condition requiring a higher dose of corticosteroid than 5 mg prednisone/prednisolone once daily
  * Active infection requiring systemic therapy
  * History of gastrointestinal disorders (medical disorders or extensive surgery) that may interfere with the absorption of the study agents
  * Uncontrolled hypertension (systolic blood pressure (BP) ≥ 160 mmHg or diastolic BP ≥ 95 mmHg); participants with a history of hypertension are allowed provided blood pressure is controlled by anti-hypertensive treatment (systolic BP <160 mmHg or diastolic BP <95 mmHg)
  * Acute or chronic hepatitis B or hepatitis C infection. (Hepatitis B and C testing are not mandatory)
* Presence of hepatitis B surface antibody is acceptable

  * Baseline moderate and severe hepatic impairment (Child Pugh Class B & C)
  * Human immunodeficiency virus (HIV)-positive participants with 1 or more of the following:
* Not receiving highly active anti-retroviral therapy.
* A change in anti-retroviral therapy within 6 months of the start of screening (except if, after consultation with the principal investigator (PI) / sponsor, a change is made to avoid a potential drug-drug interaction with the study drug).
* Receiving anti-retroviral therapy that may interfere with the study drug(s) (consult the PI / sponsor for review of medication prior to enrollment).
* CD4 count < 350 cell/mm3 at screening.
* An acquired immunodeficiency syndrome-defining opportunistic infection within 6 months of the start of screening.
* HIV testing is not mandatory

  * History of pituitary or adrenal dysfunction
  * Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) Class III or IV heart disease or cardiac ejection fraction measurement of < 50% at baseline, or clinically significant ventricular arrhythmias within 6 months prior to treatment start.
  * History of seizure or any condition that may predispose to seizure (including, but not limited to prior stroke, transient ischemic attack or loss of consciousness

    ≤1 year prior to treatment start; brain arteriovenous malformation; or intracranial masses such as schwannomas and meningiomas that are causing edema or mass effect)
  * History of an inflammatory bowel disease (Crohn's or ulcerative colitis)
  * Any additional medications that investigators are concerned will affect the response to immunotherapy.
* Use of any prohibited concomitant medications precluding safe treatment with ADT or an ARSI within 14 days prior to treatment start.

Note: Medications known to lower the seizure threshold must be discontinued or substituted at least 4 weeks prior to treatment start

* Known allergies, hypersensitivity or intolerance to apalutamide, enzalutamide, daralutamide or GNRH agonist or GNRH antagonist
* Participants that cannot tolerate MRI

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2029-03-28 (Estimated); Study Completion 2029-03-28 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a complete response or minimal residual disease. | 24 months
  To determine the proportion of patients in each cohort in whom a pathologic complete response (pCR) or minimal residual disease (pMRD, ≤ 5mm tumor) is observed in the resected primary tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Dallos, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Limited protocol activity), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All protocol activites), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activites), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org